CLINICAL TRIAL: NCT02713906
Title: Prospective Monocentric Clinical Investigation Using the Materialise X-ray Knee Guides for Total Knee Arthroplasty
Brief Title: Materialise X-ray Knee Guides for Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device not available anymore.
Sponsor: Materialise (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMAT007
Record Dates: First submitted 2015-09-25; First posted 2016-03-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Arthroplasty; Replacement; Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-Ray Knee Guide group (Experimental): Total knee arthroplasy using Materialise X-Ray Knee Guides
  Interventions: Device: X-Ray Knee Guide group

INTERVENTIONS:
Device: X-Ray Knee Guide group

SUMMARY:
The purpose of this study is to assess the positioning of customized guides designed from patients X-Rays (Materialise X-Ray Knee Guides) using computed tomography in primary total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally able and willing to comply with the protocol
* Be treated for a primary total knee arthroplasty
* Are fluent in Dutch or French
* Sign the Informed Consent Form
* Comply with the indications listed in the Instructions for Use
* Be able to undergo a CT scan

Exclusion Criteria:

* Fulfilling one of the contraindications mentioned in the Instructions for Use
* Pregnant
* A prisoner
* Reported to have mental illness or belonged to a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Difference between planned and achieved tibial and femoral components position as assessed by 3D imaging processing methods | 2 Months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Roger Jaeken, MD, Principal Investigator — AZ Heilige Familie
Locations (1):
- AZ Heilige Familie, Reet, Belgium